CLINICAL TRIAL: NCT02821182
Title: A Phase II Trial of Stereotactic Body Radiotherapy With Concurrent Anti-PD1 Treatment in Metastatic Melanoma.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: GZA Ziekenhuizen Campus Sint-Augustinus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EC UZG 2016/0540
Record Dates: First submitted 2016-06-24; First posted 2016-07-01 (Estimated); Last update posted 2022-12-29 (Actual); Status verified 2022-12

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Radiosurgery

ARMS (1):
- Anti-PD1 treatment in combination with SBRT (Experimental): Patients receiving anti-PD1 treatment will be treated with high-dose radiotherapy to one lesion in 3 fractions prior to the second cycle of systemic therapy.
  Interventions: Radiation: stereotactic body radiotherapy

INTERVENTIONS:
Radiation: stereotactic body radiotherapy — In patients with metastatic melanoma, anti-PD-1 treatment will be combined with stereotactic body radiotherapy (SBRT).
  A total dose of 24 Gy SBRT will be delivered in 3 fractions to one measurable lesion and fractions will be separated >48h and <96h.

SUMMARY:
We hypothesize that combining anti-PD1 treatment with radiotherapy might result in improved clinical response rates and PFS compared to anti-PD1 treatment in monotherapy.

The current phase II trial aims at exploring the suggested benefits of the combination and aims to improve local and distant tumour responses by exploiting the pro-immunogenic effects of radiotherapy in addition to anti-PD1 treatment.

ELIGIBILITY:
Inclusion Criteria:

* Before patient registration, written informed consent must be given according to ICH/GCP, and national/local regulations.
* Histologically confirmed diagnosis of melanoma
* At least 3 extracranial measurable metastatic lesions per RECIST v1.1. All radiology studies must be performed within 28 days prior to registration
* First line anti-PD1 treatment.
* Karnofsky Performance status > 60
* Age 18 years or older
* Female participants of childbearing potential must be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study treatment
* Female participants who are breastfeeding or plan to breastfeed should be instructed to discontinue nursing during treatment.
* Male participants must agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study treatment
* Demonstrate adequate organ function defined as the following:

  * AST and ALT ≤2.5 X ULN or ≤5 X ULN with liver metastases
  * Serum total bilirubin ≤1.5 X ULN or direct bilirubin ≤ULN for patient with total bilirubin level >1.5 ULN
  * Serum creatinine ≤1.5 X ULN
  * Absolute neutrophil count >1,000 /mcL
  * Platelets >75,000 /mcL
  * Hemoglobin >9 g/dL or > 5.6 mmol/L
* No history of active autoimmune disease requiring systemic treatment within the past 3 months or documented history of clinically severe autoimmune disease, or syndrome that requires systemic steroids or immunosuppressive agents
* Prior malignancy: Subjects who have had another malignancy should be disease-free for 5 years, or should have a history of completely resected non-melanomatous skin carcinoma or successfully treated in situ carcinoma
* No evidence of interstitial lung disease
* No uncontrolled central nervous metastases and/or carcinomatous meningitis.
* No prior radiotherapy interfering with SBRT.
* No concomitant therapy with IL-2, interferon, other immunotherapy regimens, chemotherapy, immunosuppressive agent or chronic use of systemic corticosteroids.
* No active infection requiring systemic therapy
* No known history of human immunodeficiency virus (HIV)
* No known active Hepatitis B or Hepatitis C
* Did not receive a live vaccine within 30 days prior to start of study treatment
* No mental condition rendering the patient unable to understand the nature, scope and possible consequences of the study
* Patient not unlikely to comply with the protocol; i.e. uncooperative attitude, inability to return for follow-up visits, and unlikely to complete the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2018-09-09 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Efficacy | 12 weeks
  Objective responses will be measured using RECIST v1.1. Objective responses will be defined as the number of patients with complete or partial responses as best response during follow-up.

SECONDARY OUTCOMES:
Immunologic responses | 12 weeks
  Immunologic responses will be assessed using peripheral blood samples, analyzed with FACS phenotyping, functional testing and ELISA.
  Changes in immunological parameters in tissue will be analyzed using immunohistochemistry.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Ghent, Ghent, West Vlaanderen, Belgium

REFERENCES:
- [Derived] De Wolf K, Kruse V, Sundahl N, van Gele M, Chevolet I, Speeckaert R, Brochez L, Ost P. A phase II trial of stereotactic body radiotherapy with concurrent anti-PD1 treatment in metastatic melanoma: evaluation of clinical and immunologic response. J Transl Med. 2017 Jan 31;15(1):21. doi: 10.1186/s12967-017-1123-x. PMID 28137295